CLINICAL TRIAL: NCT06638151
Title: Clopidogrel Plus Aspirin in Acute Ischemic Stroke Following Thrombectomy and/or Intravenous Thrombolysis (CoPrime): A Randomized Pilot Study
Brief Title: Clopidogrel Plus Aspirin in Acute Ischemic Stroke Following Thrombectomy and/or Intravenous Thrombolysis (CoPrime)
Acronym: CoPrime
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00140876
Record Dates: First submitted 2024-10-04; First posted 2024-10-15 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke
Keywords: intravenous thrombolysis; endovascular thrombectomy; recurrent stroke; Anti-platelet Medication; Aspirin; Clopidogrel; Acute ischemic stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin Group (Active Comparator)
  Interventions: Drug: Aspirin
- Dual Antiplatelet Group (Experimental)
  Interventions: Drug: aspirin + clopidogrel

INTERVENTIONS:
Drug: aspirin + clopidogrel — Enrolled patients with acute ischemic stroke will be randomly assigned to the clopidogrel plus aspirin group (300 mg loading dose of clopidogrel plus 160 mg aspirin on day 1; followed by clopidogrel 75 mg plus aspirin 81 mg daily from day 2-day 21, followed by aspirin 81 mg to be continued if no alternate treatment is indicated).
  Other Names: Dual antiplatelet treatment
  Arms: Dual Antiplatelet Group
Drug: Aspirin — Aspirin 81 mg once daily alone
  Arms: Aspirin Group

SUMMARY:
Stroke is a common cause of disability. The most common type of stroke, an ischemic stroke, is caused by a blood vessel in the brain getting blocked by a clot. When this happens, part of the brain is damaged because it is not getting the blood supply it needs. To treat this type of stroke, doctors give medication and/or do a procedure to remove the blockage and restore blood supply to the brain.

Unfortunately, patients who have had an ischemic stroke are at higher risk of having another ischemic stroke. This risk is highest in the first 21 days after a stroke. Currently, doctors give patients the medication aspirin every day, starting 24 hours after stroke treatment, to prevent recurrent strokes. However, some studies have shown that giving another medication, clopidogrel, in addition to aspirin, is safe and may work better than aspirin alone at preventing repeat strokes. Both aspirin and clopidogrel are a type of medication called an antiplatelet that prevents clots from forming in the blood. When both medications are given together, it is called dual antiplatelet treatment. The main risk of antiplatelet medications is bleeding.

This research aims to study the safety and feasibility of using dual antiplatelet treatment to prevent recurrent strokes. Patients who have received treatment for an ischemic stroke will first be screened to rule out patients at high risk of bleeding. Following informed consent, patients at low risk of bleeding will be enrolled in the study 24 hours after their initial stroke treatment. Patients will be randomly assigned to either take aspirin alone or aspirin and clopidogrel for 21 days for recurrent stroke prevention. The study team will then follow patients for three months after treatment to collect information about their recovery and assess differences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be >18 years of age at the time of randomization
2. Acute non-cardioembolic ischemic stroke in the anterior circulation treated with reperfusion therapy defined as intravenous thrombolysis (IVT) and/or endovascular thrombectomy (EVT)
3. Time from end of acute reperfusion therapy to randomization ≤ 24 hours
4. Mild to moderate deficit defined as a National Institute of Health stroke scale of ≤11 at the time of randomization
5. At least one non-contrast CT scan completed post reperfusion therapy and prior to randomization without any hemorrhage (including hemorrhagic infarction) and/or contrast extravasation.
6. Premorbid mRS less than or equal to 2
7. Signed informed consent from the patient or legally authorized representative

Exclusion Criteria:

1. Any known disorder associated with a significantly increased risk of bleeding
2. Post-reperfusion CT scan ASPECT score <8.
3. Anticoagulation is required for any indication other than DVT prophylaxis
4. Evidence-based indication for dual antiplatelet therapy
5. Planned surgical intervention in the next 90 days includes but is not limited to carotid endarterectomy, where dual antiplatelet is not indicated, and carotid stenting, where single antiplatelet is not used.
6. History of intracranial or subarachnoid hemorrhage
7. Intracranial tumour, arteriovenous malformation or aneurysm;
8. Intracranial or spinal cord surgery within three months;
9. Gastrointestinal or urinary tract hemorrhage within the previous 21 days;
10. Coagulation disorder, thrombocytopenia <100, 000/mm3, and Prothrombin time INR ≥1.8
11. Index stroke is caused by infective endocarditis, dissection, systematic or central nervous system vasculitis
12. History of active malignancy being treated or life expectancy ≤ 90 days
13. Allergy to clopidogrel or aspirin
14. Pregnancy
15. Participation in another clinical trial.
16. The presence of a major co-morbid illness that would make it unlikely that the participant will be able to complete follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety | 90 days
  Safety will be assessed as a proportion of patients with symptomatic hemorrhagic transformation, defined as worsening of NIHSS ≥4 compared to NIHSS at the time of randomization and hemorrhage is attributable to the antiplatelet therapy by the treatment team.
Feasibility | 21 days
  Feasibility will be assessed as a proportion of recruited patients complete the study intervention for 21 days.

SECONDARY OUTCOMES:
Early Neurological Deterioration | 7 days
  Secondary outcome measures include the proportion of patients with worsening focal neurologic deficit by NIHSS ≥4 at day seven or discharge not due to hemorrhagic transformation or any intracranial hemorrhage. Worsening will be defined as a change in NIHSS compared to NIHSS at the time of randomization.
Recurrent Stroke | 90 days
Death | 90 days
Non-Stroke Thrombotic events | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Brian Buck, Principal Investigator — University of Alberta; Mahesh Kate, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available to investigators in consultation with the principal investigators
Supporting Information: Study Protocol, ICF